CLINICAL TRIAL: NCT04831840
Title: Is PCR Amplification More Sensitive Than Urine Cultures in Diagnosing Urinary Tract Infections in Patients With Recurrent Bladder Infections?
Brief Title: Recurrent Urinary Tract Infections and the Microbiome
Status: Terminated | Type: Observational
Why Stopped: No longer with institution
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Laura Martin, Assistant Professor, University of Miami
Other Study IDs: 20201198
Record Dates: First submitted 2021-04-02; First posted 2021-04-05 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Recurrent Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female participants with recurrent urinary tract infections (RUTI).: Patients with RUTIs (Group A) will provide two urine samples. One urine sample is a clean catch and the other is a catheterized specimen. Both will be sent for analysis. A perineal swab will also be collect and analyzed for each patient.
- Female control patients without RUTIs: Patients without RUTIs (Group B) will provide two urine samples. One urine sample is a clean catch and the other is a catheterized specimen. Both will be sent for analysis. A perineal swab will also be collect and analyzed for each patient.

SUMMARY:
The primary objective is to determine if polymerase chain reaction (PCR) (UTIP™) is more sensitive in identifying urinary tract infections (UTI's) than standard urine cultures.

ELIGIBILITY:
Inclusion Criteria:

* 18 y/o-90 y/o
* Able to consent
* Female
* Group A only: Recurrent UTI (2 UTIs in 6 months)
* Group B only: No history of recurrent UTIs

Exclusion Criteria:

* Pregnant
* Pelvic radiation
* Urinary retention (>200 ml residual)
* Greater than Stage 2 prolapse
* Renal calculi
* Immunosuppressed
* Neurologic disorder with significant bladder impairment
* No current UTI via dip stick

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients with RUTIs and controls will be enrolled from University of Miami's or Holy Cross Hospital's female pelvic medicine and reconstructive surgery clinics.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Proportion of uropathogens | Day 1
  The proportion of uropathogens found on PCR versus urine culture from urine samples.
Proportion of patients negative for repeat testing | Up to 4 weeks
  The proportion of negative patient on repeat testing of urine samples.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Martin, DO, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: No